CLINICAL TRIAL: NCT03538431
Title: Improving Driving in Young People With Autism Spectrum Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Programs in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2018-P-000900
Record Dates: First submitted 2018-05-14; First posted 2018-05-29 (Actual); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; ASD; Anxiety
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders | interventions — Buspirone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Buspirone (Experimental): These subjects will receive buspirone prior to engaging in the driving simulation.
  Interventions: Drug: Buspirone
- Unmedicated (Experimental): These subjects will take no medication prior to engaging in the driving simulation
  Interventions: Drug: Buspirone

INTERVENTIONS:
Drug: Buspirone — Buspirone is an atypical anxiolytic medication.

SUMMARY:
This study will examine the effects of treatment with the anti-anxiety medicine buspirone on driving performance (eye tracking) in individuals with high-functioning autism spectrum disorder (HF-ASD).

The study consists of an Assessment Visit at Massachusetts General Hospital (MGH), as well as two Driving Simulation visits that will take place at Massachusetts Institute of Technology (MIT). Subjects will be given buspirone and asked to take the medication for the two days preceding the Driving Simulation Visit.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 18-24, with a diagnosis of DSM-V Autism Spectrum Disorder
* Has a valid Driver's License

Exclusion Criteria:

* Major sensorimotor handicaps (e.g. deafness, blindness)
* Individuals who have never held a valid driver's license
* Intellectual Deficiency (Verbal Comprehension Index < 80)
* Inadequate command of the English language
* Subjects with any clinically meaningful medical or psychiatric condition as determined by the investigator
* Individuals who are currently taking a monoamine oxidase inhibitor (MAOI) for any reason
* Pregnant

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Buspirone Before Simulation 1, Then no Buspirone Before Simulation 2: These subjects will receive and be instructed to take the buspirone for the 2 days preceding their first driving simulation visit. They will not take buspirone before their 2nd driving simulation visit.
  Buspirone: Buspirone is an atypical anxiolytic medication.
- No Buspirone Before Simulation 1, Then Buspirone Before Simulation 2: These subjects will receive and be instructed to take the buspirone for the 2 days preceding their second driving simulation visit. They will not take buspirone before their 1st driving simulation visit.
  Buspirone: Buspirone is an atypical anxiolytic medication.
Period: Overall Study
Arm/Group | Buspirone Before Simulation 1, Then no Buspirone Before Simulation 2 | No Buspirone Before Simulation 1, Then Buspirone Before Simulation 2
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Buspirone: These participants took buspirone either before driving simulation 1 or before driving simulation 2. Those who took the medication before driving simulation visit 1 took no medication before visit 2, and those who took the medication before driving simulation visit 2 took no medication before driving simulation 1. This study is a crossover design.
Arm/Group | Buspirone
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Driving Performance - Measured by Mean Off-Road Glance Duration
Description: Driving performance will be analyzed using eye tracking in individuals with Autism Spectrum Disorder while on the anti-anxiety medication buspirone and while not on buspirone. Eye movement behavior (measured by glance duration) during the driving simulation was manually coded on a frame-by-frame basis from recorded video by trained coders for all cases where usable video recordings were available for both the medicated and non-medicated driving simulation sessions per participant.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Buspirone: Subjects will receive buspirone before 1 of 2 driving simulation visits. Half of the participants in the study completed Simulation 1 on buspirone, and the other half completed Simulation 2 on buspirone. These participants completed the driving simulation on buspirone.
  Buspirone: Buspirone is an atypical anxiolytic medication.
- Unmedicated: These participants completed the driving simulation unmedicated.
  Subjects will receive buspirone before 1 of 2 driving simulation visits. Half of the participants in the study completed Simulation 1 on unmedicated, and the other half completed Simulation 2 on unmedicated.
  Buspirone: Buspirone is an atypical anxiolytic medication.
Arm/Group | Buspirone | Unmedicated
Number analyzed (Participants) | 21 | 21
Seconds | 0.85 (0.17) | 0.90 (0.27)

2. Primary Outcome: Heart Rate
Description: Hyperarousal will be measured by heart rate during participants' time in the driving simulation.
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: Beats Per Minute
Groups:
- Buspirone: These participants completed the driving simulation on buspirone.
  Subjects will receive buspirone before 1 of 2 driving simulation visits. Half of the participants in the study completed Simulation 1 on buspirone, and the other half completed Simulation 2 on buspirone.
  Buspirone: Buspirone is an atypical anxiolytic medication.
- Unmedicated: These participants completed the driving simulation without buspirone.
  Subjects will receive buspirone before 1 of 2 driving simulation visits. Half of the participants in the study completed Simulation 1 unmedicated, and the other half completed Simulation 2 unmedicated.
  Buspirone: Buspirone is an atypical anxiolytic medication.
Arm/Group | Buspirone | Unmedicated
Number analyzed (Participants) | 24 | 24
Beats Per Minute | 81.78 (10.67) | 82.74 (11.70)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant between the date the participant enrolled in the study and the date the participant completed the study. The precise time frame of this window differed by participant depending on their availability to schedule the driving simulations. On average, adverse event data were collected over a period of 7.2 weeks.
Groups:
- Buspirone: These subjects received buspirone either before driving simulation visit 1 or before driving simulation 2.
- Unmedicated: These subjects received no medication either before driving simulation visit 1 or before driving simulation 2.
Arm/Group | Buspirone | Unmedicated
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 5/26 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone (N=26) | Unmedicated (N=26)
Mild allergic reaction to medication prescribed not related to the study (Immune system disorders) | 1 (1) | 0 (0) — The participant reported having a mild allergic reaction to vitamins B12 and D3 that were prescribed by the primary care physician. This was determined to be unrelated to the study drug.
Concussion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The subject reported receiving a concussion between enrolling in the study and medication driving simulation visit. The concussion healed prior to the drive. This was determined to be unrelated to the study
Chest Tightness, mild excitement, and nausea (Cardiac disorders) | 1 (1) | 0 (0) — Participant reported suffering from chest tightness, mild excitement, and nausea while taking the new medication. Chest tightness was possibly related, and excitement and nausea were related to the drug. All resolved 24 hours after onset.
Mild nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant endorsed nausea as a side effect of buspirone medication. This side effect was mild, expected, and related to the study drug. It resolved 24 hours after onset.
Head Cold (Infections and infestations) | 1 (1) | 0 (0) — The subject reported having a head cold during the medication driving simulation visit and was not able to sleep. This event was considered mild and unrelated to the study drug,

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT03538431/Prot_SAP_001.pdf